CLINICAL TRIAL: NCT00002988
Title: Phase I Treatment of Adults With Primary Malignant Glioma With Irinotecan (CPT-11) (NSC #6616348) Plus BCNU (NSC #409962)
Brief Title: Irinotecan Plus Carmustine in Treating Patients With Recurrent Primary Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 0564; DUMC-000564-00-3R3; DUMC-0509-99-3R2; DUMC-0509-99-4R1; DUMC-427-98-3R1; DUMC-461-97-3; NCI-G97-1243; CDR0000065523 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-05-19 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — Carmustine; Irinotecan

INTERVENTIONS:
Drug: carmustine
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of irinotecan plus carmustine in treating patients who have recurrent primary malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of irinotecan administered in combination with a fixed dose of carmustine in patients with recurrent primary malignant glioma. II. Determine the toxic effects of irinotecan and carmustine in these patients.

OUTLINE: This is a dose escalation study of irinotecan. Patients receive irinotecan IV over 90 minutes weekly on weeks 1-4 and carmustine IV over 1 hour on weeks 1-6. Treatment continues in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose limiting toxicities.

PROJECTED ACCRUAL: Approximately 18-36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent primary malignant glioma Measurable recurrent or residual primary central nervous system neoplasm confirmed by MRI

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: Karnofsky 60-100% Hematopoietic: Hematocrit greater than 29% Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 125,000/mm3 Hepatic: SGOT less than 1.5 times upper limit of normal (ULN) Bilirubin less than 1.5 times ULN Renal: Creatinine less than 1.5 mg/dL BUN less than 25 mg/dL Pulmonary: DLCO at least 60% Other: Not pregnant Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 6 weeks since prior chemotherapy No prior irinotecan or carmustine treatment failure No more than 1 prior chemotherapy regimen Endocrine therapy: Patients taking corticosteroids must be on a stable dose for at least 1 week prior to study and the dose should not escalate over entry dose level Radiotherapy: At least 6 weeks since prior radiotherapy Surgery: At least 3 weeks since prior surgical resection Other: No concurrent medication that may interfere with study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 1997-04; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States